CLINICAL TRIAL: NCT06460350
Title: Enhancing Pain Management for Knee Replacement Patients Through an Innovative Non-invasive and Opioid-sparing Device (NEUROCUPLE™)
Brief Title: NEUROCUPLE™ in TKA Patients to Enhance Pain Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: nCap Medical (Industry)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY24020075
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Total Knee Arthroplasty

STUDY DESIGN:
Intervention Model Description: This will be a double-blinded randomized (1:1) placebo-controlled clinical trial to determine the feasibility and effectiveness of a 2-week application of the NEUROCUPLE device for pain relief and reduction of opioid refills after TKA. We have a placebo device (sham device without the captor array layer) that looks exactly like the active device, allowing us to conduct a true placebo-controlled randomized study. The trial will include 140 participants over a 1-year period.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- NEUROCUPLE™ Group (Experimental): This arm of subjects will receive the active NEUROCUPLE™ patch to wear for 2-weeks following their TKA surgery.
  Interventions: Device: NEUROCUPLE™ Patch
- Placebo Group (Placebo Comparator): This arm of subjects will receive the placebo (non-active, sham) patch to wear for 2-weeks following their TKA surgery.
  Interventions: Device: Placebo Patch

INTERVENTIONS:
Device: NEUROCUPLE™ Patch — nCAP Medical has developed an effective, safe, non-opioid alternative, the NEUROCUPLE™ device, based on an innovative nanotechnology to reduce surgical pain and facilitate functional recovery while reducing opioid prescriptions, opioid-related adverse events and reducing the cost of care in millions of Americans undergoing TKA each year.
  Arms: NEUROCUPLE™ Group
Device: Placebo Patch — The placebo patch is identical to the active patch but with no active agents.
  Arms: Placebo Group

SUMMARY:
This is a randomized (1:1) placebo-controlled clinical trial to determine the feasibility and effectiveness of 30-day application of NEUROCUPLE™ patch for pain reduction and opioid consumption following TKA. Results will establish NEUROCUPLE™ as an effective non-opioid postoperative pain management device for FDA approval. Importantly, we have a placebo device (device without the captor array layer) that looks exactly like the active device, allowing us to conduct a true placebo randomized study.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is the most common elective surgical procedure. By 2030, 3.5 million TKA procedures are expected1 to be performed. Multiple factors can contribute to an individual's need for TKA; however, the primary factor is osteoarthritis15 and pain. Osteoarthritis affects approximately 32.5 million individuals in the US, leading to an enormous economic burden, ranging from $15-$16 billion dollars annually. Although most diagnosed with osteoarthritis should undergo TKA, the fear of experiencing severe long lasting postoperative pain causes many to postpone the surgery. For those that do elect surgery, postoperative pain decreases quality of life and an increase in risk of chronic opioid use. Out of 98,623 individuals who received TKA from 2015 to 2019, it was reported that 72% received opioid prescriptions in duration and dosage, which was proposed to be the cause of long-term opioid use.

Postoperative pain strategies for TKA often requires opioid use. To mitigate postoperative pain management following TKA a multimodal approach is often used as a part of enhanced recovery after surgery (ERAS) protocols. This approach on the use of on peripheral nerve blocks (PNB)s, acetaminophen, non-steroidal anti-inflammatory drugs (NSAIDs), and opioids13,18,19. Postoperative opioid and NSAIDS can lead to excessive sedation, vomiting, nausea, hypotension, major bleeding, life-threatening respiratory depression, constipation, renal failure, frequent delayed functional recovery, increase cost of care, and prolong hospital stay. Furthermore, the postoperative prescription of use opioids leads to long-term opioid users in 34.7% to 53.5%. Patients with poorly controlled acute surgical pain are at risk for chronic post-surgical pain, opioid dependence, and long-term opioid use. Thus, there is an urgent and unmet clinical need for a reliable technology to predict and reduce opioid use and costly opioid adverse effects while enhancing surgical pain relief. On an economic point of view, evidence also demonstrates that persistent postoperative pain leads to a loss in work productivity and absenteeism, mounting to an average loss of $13,761 per individual. Therefore, there is a significant need for alternative non-pharmacological, and non-opioid therapies that are effective in treating postoperative pain management in patients undergoing TKA.

Clinical approaches associated with postoperative pain and opioids in TKA. Data compiled from 90 million patients from 38 hospital networks and 18 non-network hospitals demonstrated that reliance on opioids for postoperative pain management is still extremely high (91.5%) following a TKA. Evidence supporting the use of PNBs is lacking and their use may increase the risk of fall. Sharma et al., 2010 reported that femoral nerve blocks conducted in 709 patients lead to postoperative falls (n=13 patients). A study including 250 patients demonstrated that postoperative falls led to an extended hospital stay. Furthermore, nerve injury and major bleeding have also been reported following PNBs. Complementary techniques such as Transcutaneous Electrical Nerve Stimulation (TENS), acupuncture and hypnosis have been proposed but evidence supporting the use of these techniques is still limited and the use of these techniques requires expertise and time. Therefore, current postoperative pain treatments remain unsatisfactory.

A pain relief patch that provides a clinically effective alternative to opioid use for pain management. The scientific premise of our proposal rests upon the published literature and our preliminary data that demonstrates the use of pain relief patches for pain management. Pain and local inflammation following tissue injuries is the result of the release of a number of mediators and ions, decreases in pH (increase in acidity), and changes in local electrical potential. This is in part due to the central nervous system stimulation of nociceptors and the anterior and lateral spinothalamic tracts. The NEUROCUPLE™ device's millions of nanocapacitors capture and release the excess electrical load generated by trauma, thus blocking the transmission of the local pain signals.

An observational study evaluating non-surgical patients' (n=66) using our licensed nanotechnology topical analgesic demonstrated a 71% reduction in Brief Pain Inventory pain severity (Fig. 1), improvements in quality of life, and a 98% reduction in oral pain medication use. Our additional preliminary data in patients undergoing a TKA demonstrated that the use of the patch device plus standard on care was associated with a 36% reduction in pain at rest by postoperative day 3 and more importantly a reduction of 47% in the number of patients requesting an opioid refill beyond their initial prescription within the first 30 days compared to the patients receiving only standard of care. Thus, we believe our clinical data provides a strong scientific premise for utilizing pain relief patches as an alternative to analgesic drugs to provide effective and safe postoperative approach to reduce postoperative analgesia and more importantly to greatly reduce the number of patients requiring long term opioid exposure which has been demonstrated as a risk for postoperative opioid use disorder (OUD) in surgical patients.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Scheduled for elective primary unilateral TKA
* T-score < 60 on the PROMIS Anxiety measure

Exclusion Criteria:

* Children (<18 yr.)
* Pregnant women
* Active alcoholism (defined as daily use of more than 1 liter of wine and /or 3 or more shots of hard liquor) or drug abuse (defined as daily use of illicit drugs)
* Severe chronic pain condition that requires daily preoperative opioid dependence
* T-score ≥ 60 in any of the three PROMIS measures (i.e., sleep, anxiety, and depression)
* Other concomitant surgery being performed in addition to TKA
* Patients undergoing bilateral TKA
* Patients undergoing knee replacement revision
* Patients with limited mobility (in a wheelchair or requiring a walker)
* Patients who are not returning home after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2024-09-25 (Actual); Primary Completion 2025-07-18 (Actual); Study Completion 2025-07-18 (Actual)

PRIMARY OUTCOMES:
Post-operative pain at rest | 1-Week Post Hospital Discharge
  Pain at rest will be assessed by a numerical rate scale (NRS), in which 0 = no pain at all and 10 = the worst pain imaginable

SECONDARY OUTCOMES:
Post-Operative Nausea and Vomiting | Up to 24-hours post-operatively
  Incidence of PONV measured by antiemetic use yes/no
Time to hospital discharge (length of hospital stay) | Up to post-operative day 7
  The length of the hospital stay will be abstracted from the medical records and the averaged time [mean(SD)] will be reported in minutes.
Total Opioid Use in OME (mg) (in hospital) | Up to 24-hours post-operatively
  OME measured in mg
Total Opioid Use in OME (mg) at 1 week | One-week Post Hospital Discharge
  OME measured in mg
Post-Operative pain scores (NRS) | Up to 24-hours post-operatively
  Assessed by a numerical rate scale (NRS), in which 0 = no pain at all and 10 = the worst pain imaginable

OTHER OUTCOMES:
Baseline pain at rest | Prior to day of surgery
  Pain at rest will be assessed by a numerical rate scale (NRS), in which 0 = no pain at all and 10 = the worst pain imaginable
Pain while walking 30 feet, baseline | Prior to day of surgery
  Pain while walking 30 feet will be assessed by a numerical rate scale (NRS), in which 0 = no pain at all and 10 = the worst pain imaginable
Pain while walking 30 feet, 1-week post-op | 1-Week Post Hospital Discharge
  Pain while walking 30 feet will be assessed by a numerical rate scale (NRS), in which 0 = no pain at all and 10 = the worst pain imaginable
Pain while walking 30 feet, 6-weeks post-op | 6-Weeks Post Hospital Discharge
  Pain while walking 30 feet will be assessed by a numerical rate scale (NRS), in which 0 = no pain at all and 10 = the worst pain imaginable
Pain while walking 100 feet, baseline | Prior to day of surgery
  Pain while walking 100 feet will be assessed by a numerical rate scale (NRS), in which 0 = no pain at all and 10 = the worst pain imaginable
Pain while walking 30 feet, 2-weeks post-op | 2-Weeks Post Hospital Discharge
  Pain while walking 30 feet will be assessed by a numerical rate scale (NRS), in which 0 = no pain at all and 10 = the worst pain imaginable
Pain while walking 100 feet, 1-week post-op | 1-Week Post Hospital Discharge
  Pain while walking 100 feet will be assessed by a numerical rate scale (NRS), in which 0 = no pain at all and 10 = the worst pain imaginable
Pain while walking 100 feet, 2-weeks post-op | 2-Weeks Post Hospital Discharge
  Pain while walking 100 feet will be assessed by a numerical rate scale (NRS), in which 0 = no pain at all and 10 = the worst pain imaginable
Pain while walking 100 feet, 6-weeks post-op | 6-Weeks Post Hospital Discharge
  Pain while walking 100 feet will be assessed by a numerical rate scale (NRS), in which 0 = no pain at all and 10 = the worst pain imaginable
Opioid prescriptions within the first 6-weeks following surgery | 6-Weeks Post Hospital Discharge
  The number of opioid refills will be collected via Prescription Drug Monitoring Program (PDMP) for up to 6-weeks following hospital discharge. This will be averaged across each group and reported as a Mean(SD).
Patient Satisfaction with overall care | 2-Weeks and 6-Weeks Post Hospital Discharge
  Scale from 0 (least satisfied) to 10 (most satisfied)
Patient Satisfaction with pain management | 2-Weeks and 6-Weeks Post Hospital Discharge
  Scale from 0 (least satisfied) to 10 (most satisfied)
Pain while walking 100 feet, 24-hours post-op | 24-hours post-operatively
  Pain while walking 100 feet will be assessed by a numerical rate scale (NRS), in which 0 = no pain at all and 10 = the worst pain imaginable
Pain while walking 30 feet, 24-hours post-op | 24-hours post-operatively
  Pain while walking 30 feet will be assessed by a numerical rate scale (NRS), in which 0 = no pain at all and 10 = the worst pain imaginable

CONTACTS AND LOCATIONS:
Overall Officials: Jacques E. Chelly, MD, PhD, MBA, Principal Investigator — University of Pittsburgh / UPMC
Locations (1):
- UPMC Shadyside Hospital, Pittsburgh, Pennsylvania, United States